CLINICAL TRIAL: NCT04910451
Title: Investigating the Safety and Effect of Overnight Orthokeratology and Its Influencing Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-448
Record Dates: First submitted 2021-05-31; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Myopia
Keywords: orthokeratology; myopia control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention

SUMMARY:
To investigate the Safety and Effect of Overnight Orthokeratology and Its Influencing Factors in China

DETAILED DESCRIPTION:
Patients who were successfully prescribed with orthokeratology lenses in Eye Center of the Second Affiliated Hospital of Zhejiang University School of Medicine were enrolled in the study. Our study used two different methods to collect data. For complications and effect of orthokeratology information, data were collected by a retrospective survey. A questionnaire was used to collect influencing factors of safety and effect of orthokeratology.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were successfully prescribed with ortho-k lenses in Eye Center of the Second Affiliated Hospital of Zhejiang University School of Medicine

Exclusion Criteria:

* Patients who have ceased wearing orthokeratology or who were using other methods of myopia control

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: myopia patients who were using orthokeratology for myopia control
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
axial length | 1 year
  changes in axial length

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwen Bian, doctor, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China